CLINICAL TRIAL: NCT03228446
Title: Improving Cognitive Functions by Training Distractor Inhibition (DIIN) in Younger and Older Healthy Adults
Brief Title: The Effects of Attentional Filter Training on Working Memory
Acronym: DIIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Notger Müller, Prof. Dr. med. (Head of Neuroprotection Lab at the DZNE), German Center for Neurodegenerative Diseases (DZNE)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD021
Record Dates: First submitted 2017-07-12; First posted 2017-07-25 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Decline; Healthy; Age-related Cognitive Decline
Keywords: training intervention; filter training; distractor inhibition
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young subjects (Experimental): Working memory training & attentional filter training for participants (18-30 years)
  Interventions: Behavioral: filter training; Behavioral: memory training
- Old subjects (Experimental): Working memory training, attentional filter training and no training (control) for participants (60-80 years)
  Interventions: Behavioral: filter training; Behavioral: memory training; Other: no training (control)

INTERVENTIONS:
Behavioral: filter training — one-week filter training on the computer: computerized visual change detection experiment (selective attention )
Behavioral: memory training — one-week storage training on the computer: computerized visual change detection experiment (memory storage)
Other: no training (control) — no training applied
  Arms: Old subjects

SUMMARY:
The investigators are interested in how attentional filter training/ distractor inhibition training could influence cognitive functions like working memory, executive control, problem solving, decision making and attentional control.

DETAILED DESCRIPTION:
Two different computer based trainings were applied: an attentional filter training and a working memory training.

ELIGIBILITY:
Inclusion Criteria:

* right-hander
* aged between 18-30 or 60-80years

Exclusion Criteria:

* severe visual impairments (e.g. dyschromatopsia, very low vision)
* diseases or medication that might impair test performance
* Montreal Cognitive Assessment Score (MoCA) < 26 points

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09-26 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Improvements in test performance | 45min pre / post
  Working memory and filtering performance (in %), effects of distractor interference and reaction times for trials with and without distractors with 4, 5 & 6 targets

SECONDARY OUTCOMES:
Rey Complex Figure Test | 30min pre / post
  Copying complex figures and reproduce it from memory
Memory from TAP (Test battery of Attentional Performance) | 45min pre / post
  Working Memory (n-back)
Attention from TAP (Test battery of Attentional Performance) | 45min pre / post
  divided attention, Go-NoGo, Flexibility, Incompatibility, Visual scanning
Performance in repeating numbers | 10min pre / post
  Repeating numbers in forward & backward conditions
Subtest from CANTAB (Cambridge Neuropsychological Test Automated Battery) | 10min pre / post
  Spatial Span Test
Iowa Gambling Task | 5min on each training day (1-5)
  Decision making
Daily Questionnaires | 2 min on each training day (1-5)
  subjective performance in the training paradigm
Daily Questionnaires | 2min on each training day (1-5)
  Assessing external circumstances of daily influences
Memory performance without distractors among different setsizes | 45min pre / post
  Working memory performance (in %) for trials with 4, 5 & 6 targets and averaged performance for all conditions without distractors
Memory performance with distractors among different setsizes | 45min pre / post
  Working memory performance (in %) for trials with 4, 5 & 6 targets and distractors and averaged performance for all conditions with distractors
Filtering performance without distractors among different setsizes | 45min pre / post
  Filtering performance (in %) for trials with 4, 5 & 6 targets and averaged performance for all conditions without distractors
Filtering performance with distractors among different setsizes | 45min pre / post
  Filtering performance (in %) for trials with 4, 5 & 6 targets and distractors and averaged performance for all conditions with distractors
Reaction times | 45min pre / post
  Reaction times in each condition
Values of distractor inhibition | 45min pre / post
  Distractor inhibition (DIIN) = Mean of conditions without distractors - Mean of conditions with distractors

CONTACTS AND LOCATIONS:
Overall Officials: Notger Müller, Prof. Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (1):
- DZNE, Magdeburg, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmicker M, Schwefel M, Vellage AK, Muller NG. Training of Attentional Filtering, but Not of Memory Storage, Enhances Working Memory Efficiency by Strengthening the Neuronal Gatekeeper Network. J Cogn Neurosci. 2016 Apr;28(4):636-42. doi: 10.1162/jocn_a_00922. Epub 2016 Jan 14. PMID 26765946
- [Result] Schmicker M, Muller P, Schwefel M, Muller NG. Attentional Filter Training but Not Memory Training Improves Decision-Making. Front Hum Neurosci. 2017 Mar 23;11:138. doi: 10.3389/fnhum.2017.00138. eCollection 2017. PMID 28386225